A Phase I Single-Arm Open Label Dose-Escalation Study of CivaSheet With Radical Prostatectomy With or Without Adjuvant External Beam Radiation Therapy in Patients With High Risk Prostate Cancer

Dr. Ketan Badani NCT03657108

Document Date: 10-18-2022

**** 

| <b>Study ID</b> : 16-1314 | Form Version Date: 6/29/2021 |
|---|---|
| STUDY INFORMATION: | |
| • | Open Label Dose-Escalation Study of CivaSheet with Radica<br>vant External Beam Radiation Therapy in Patients with High Ris |
| Principal Investigator (Head Rese | archer): Ketan Badani, MD |
| <b>Physical Address:</b> Mount Sinai We 10019 | st Hospital: , New York, N |
| Mailing Address: | , New York, NY 10019 |
| <b>Phone:</b> 212-241-3919 | |

#### SUMMARY OF THIS RESEARCH STUDY:

In medicine there are many unanswered questions. A research study is when scientists try to answer a question about something that we don't know enough about. Participation in a research study may or may not directly help you or others. Participation is entirely voluntary. It is completely up to you whether or not you take part. You can also change your mind at any time and it will not affect your ability to get medical care within the Mount Sinai Health System.

The purpose of this study is to determine whether CivaSheet® combined with radical prostatectomy and external beam radiation is safe as a treatment for high risk prostate cancer. CivaSheet® has never been used in the treatment of high risk prostate cancer. Therefore, the purpose of this study is also to determine the highest dose of the CivaSheet® not yielding unacceptable toxicity (the amount of damage caused by the CivaSheet®).

If you choose to participate:

- You would agree to undergo study procedures including follow-up visits, imaging, radical prostatectomy with permanent CivaSheet® implant and external beam radiation therapy.
- You would agree to fill out questionnaires before surgery and at each follow up visit after surgery requiring these questionnaires to be filled out
- You would agree to share relevant follow up clinical information when asked via mail or telephone for duration of 5 years after enrollment in the study.

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. While we hope that CivaSheet® with Radical Prostatectomy and Adjuvant External Beam Radiation Therapy will result in a reduced risk of cancer spread, a reduced risk of cancer




**Study ID**: 16-1314 **Form Version Date: 6/29/2021** 

recurrence and a reduced risk of death from prostate cancer, there is no evidence that this will occur. While we also hope that this combination treatment will reduce the unfavorable genitourinary and gastrointestinal effects of radiation to the bladder and rectum, there is no evidence that this will occur. Results from this trial may result in benefits to others. Determining the best dose of the CivaSheet® and whether this combination treatment is safe in this trial will allow us to safely treat future patients with the best dose of the CivaSheet® combined with radical prostatectomy and external beam radiation therapy to potentially reduce the risk of cancer spread, recurrence, death and complications related to radiation in other patients

If you are interested in learning more about this study, please continue to read below.

#### PARTICIPATION IN THIS RESEARCH STUDY:

This research study will be fully explained to you by a member of the study team. Feel free to ask all the questions you want before you make a decision about whether or not to participate. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

You may qualify to take part in this research study because you have prostate cancer, are eligible for radical prostatectomy and external beam radiation therapy and fall into one of the following categories:

- Category 1:
  - One of the following features present:
    - Clinical stage ≥T3a, Gleason score ≥ 8, or PSA > 20
- Category 2:
  - One of the features present from both categories 2a and 2b:
    - Category 2a: Clinical stage T2b, Clinical stage T2c, Gleason score 7, or PSA 10-20.
    - Category 2b: Seminal vesicle invasion, Extracapsular extension, or Lymph node positive disease.

Funds for conducting this research are provided by Civatech Oncology, Inc. This company manufactures the CivaSheet® and specializes in the production of low dose rate brachytherapy products.

#### LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE:

Your participation in this research study is expected to last 10 months.

This is a multisite study. The number of people expected to take part in this research study at Mount Sinai Hospital is 4. The number of people expected to take part in this research study at Mount Sinai West Hospital is 4. The number of people expected to take part in this research study at Mount Sinai St. Luke's hospital is 4. The total number of people expected to take part in this research study is 12.



**** 


#### **DESCRIPTION OF WHAT'S INVOLVED:**

If you agree to participate in this research study, the following information describes what may be involved.

- Research activities will take place at Mount Sinai Hospital, Mount Sinai West Hospital and Mount Sinai St. Luke's Hospital. You can choose to go to more than one of the locations for different study visits.
- If you take part in this study, you will have the following tests and procedures:
  - Consent to participation in this study. Educational materials will be provided and all aspects of the study design, risks, benefits, procedures and responsibilities of the patient will be discussed.
  - 2. Review of eligibility criteria to determine if you are eligible for participation in this study.
  - 3. **Pre-operative Visit:** A visit to document your medical history, current medications, baseline sexual and urinary function, and adverse event history.
    - a. Completion of three questionnaires.
      - i. International Index of Erectile Function Questionnaire: A questionnaire evaluating sexual function: Completion of this questionnaire takes 5-10 minutes.
    - b. Assessment of baseline physical status.
    - c. Scheduling of standard of care radical prostatectomy and experimental procedure Civasheet® implant.
    - d. The length of this visit will be approximately 1 hour long.

#### 4. Experimental Procedures:

- a. After your pre-operative visit and medical clearance is obtained: You will undergo standard of care radical prostatectomy and the experimental device CivaSheet® will be permanently placed inside of you during the surgery. Based on our identification of areas where cancer is likely to be left behind and areas that are suspicious for cancer spread based on your pre-operative MRI, CivaSheet® will be permanently placed and sewn onto these areas during your surgery to remove the prostate.
- b. Radical prostatectomy is a procedure to remove the prostate and surrounding tissue and is part of regular medical care for your prostate cancer which will be done even if you decide to not take part in the research.
- c. The length of this procedure will be 3-4 hours long. In total, you should plan to be in the hospital for 2-3 days.



#### 

**Study ID**: 16-1314

5. One month after your surgery to remove the prostate and implantation of the CivaSheet®: You will receive a computed tomography (CT) so that your doctor can assess exactly where the radiation will be aimed during external beam radiation. The length of this procedure will be 1 hour.

Form Version Date: 6/29/2021

- 6. Six weeks after your surgery to remove the prostate and implantation of the CivaSheet®: You will receive standard of care external beam radiation every day from Monday to Friday for 5 weeks to your pelvic area (the region of your body between your abdomen and thighs).
  - a. External beam radiation therapy following radical prostatectomy is a procedure consisting of delivery of high-energy x-rays to cancerous areas surrounding the prostate and is part of regular medical care for your high risks prostate cancer which will be done even if you decide to not take part in the research.
  - b. This procedure will take 30-60 minutes every day from Monday to Friday for 5 weeks.
- 7. **3 months after removal of the prostate and implant of the CivaSheet**<sup>®</sup>: you will receive a computed tomography (CT) scan to assess whether the CivaSheet<sup>®</sup> is still in place. The length of this procedure will be 1 hour.
- **8. Follow-Up Tests and Procedures:** These visits are part of the regular medical care for advanced prostate cancer which will be done even if you decide to not take part in the research.
  - a. Frequency of Follow-Up Visits:
    - i. 1 week after removal of the prostate and implant of the CivaSheet<sup>®</sup>.
    - ii. 6 weeks, 3 months and 6 months after External Beam Radiation Therapy.
    - iii. Yearly routine follow-up per standard of care for 4 years.
  - b. Length of Follow-up
    - i. The length of each visit will be 15-30 minutes
  - c. Procedures at Follow-Up Visits:
    - i. Completion of the Health Related Quality of Life Questionnaire
    - ii. Completion of the International Index of Erectile Function Questionnaire
    - iii. Expanded Prostate Cancer Index Composite (EPIC) questionnaire: A questionnaire to evaluate patient function and bother after radical prostatectomy. Takes 10 minutes to complete
    - iv. Blood Test to measure PSA (a value to determine whether your cancer has returned) and testosterone. 3 vials of blood will be drawn.



#### 


- You may be contacted by the research team for more information relating to the research during your follow up visits for routine clinical care and also via email or phone when in person visits are not feasible.
- Throughout this study, you will interact with nurses, study coordinators, the Principal Investigator, physicians at Mount Sinai Hospital sites.
- The researchers would like to ask your permission to keep data collected from you during this study to use them in future research studies. These data include your demographics (name, age, social security number, medical record number), study information (subject study ID), medical history (Other illnesses, medications, prior surgery), physical examination information (Whole body physical exam including related to the rectal exam for prostate cancer screening) information related to prostate cancer (pathology from biopsy and surgery), any imaging data pertaining to prostate cancer (CT, MRI, ultrasound, bone scan), blood tests done as part of cancer work up (PSA, testosterone - total and free), procedural data (prostatectomy, external beam radiation therapy), and responses to all study related questionnaires (for example, the International index of erectile function questionnaire, etc.) completed by subjects as part of this study. They would also like to know your wishes about how they might use your data in future research studies. You should also know that it is possible that products may someday be developed with the help of your data, and there are no plans to share any profits from such products with you. Your clinical data will be directly linked to your identifiable information (name, date of birth, medical record number, social security number). Data will be stored and maintained on a secure web application used to create and manage online clinical databases on a limited access Mount Sinai IT maintained network. This application called Research Electronic Data Capture (REDCap) allows auditing and tracking of many activities of researchers using the application to ensure that all data is accessed and used according to institutional review board regulations. All identifiable information not stored on a limited access Mount Sinai IT maintained network will be encrypted and password protected. The Principal investigator (Dr. Ketan Badani) is responsible for receipt or transmission of the data. All research team members listed on this protocol will have access to the data with identifiable data during the conduct of the trial. Data will be transmitted for use only on REDCap which is password protected and access given only to research personnel listed on this protocol.

The researchers would like to ask your permission to keep the data and specimens (like blood, tissue, hair, or any other body matter) collected from you during this study to use them in future research studies. Please tell us how we may use this material in future research studies.

| (1) Will you allow the researchers to store your information and/or specimens to use in future research studies? | | |
|---|---|---|
| Yes<br>next question. | No | If no, please stop here. If yes, please continue to the |

(2) The researchers can keep your information and/or specimens stored in one of two different ways: one way will store your information and/or specimens in a way that it is linked to your identity (through



### 

Form Version Date: 6/29/2021

| the use of a code that can indicate the information came from you personally) and the other way will store your information and/or specimens anonymously (no one will know who the information is from It will not be stored both ways, so you must choose one of these two options. Please note that if you choose to have your information and/or specimens stored anonymously, you will not be able to change your mind to ask for your information and/or specimens to be destroyed at a future date. How would you like your information and/or specimens stored? Please initial <b>ONE</b> choice: | |
|---|---|
| | formation and/or specimens stored with a link to my identity<br>formation and/or specimens stored anonymously |
| additional informa | ne researchers permission to <b>contact you</b> in the future to collect ation about you, discuss how your information and/or specimens might be used, or to participation in another research project? Please initial your choice: |
| Yes N | 0 |
| | ne researchers permission to keep the information and/or specimens indefinitely and re studies that are <b>directly related</b> to the purpose of the current study? rehoice: |
| Yes N | 0 |
| use them for futur | ne researchers permission to keep the information and/or specimens indefinitely and re studies that are <b>not related</b> to the purpose of the current study (for ent area of research)? Please initial your choice: |
| Yes N | o |
| information. This patterns etc. Do | o time researchers outside of medicine and related sciences would like to use this might be in the field of anthropology, human origins, mapping human migration you give permission to use your information and/or specimens outside the fields of logical sciences? Please initial your choice: |
| Yes N | 0 |
| the information ar <b>(b)</b> If the future re | esearch in a different area can be done without having to know that and/or specimens came from you personally, that will be done. Esearch in a different area requires that it is known specifically who the information is came from, then one of the following will be done: |

(i) If you allowed the researchers to contact you in the future, they may be able to contact you to explain why your identifiable information or specimen is needed and what will be done with it. Your

permission will be asked to use your information and/or specimens in that research project.



Effective Date: 10/18/2022 End Date:10/17/2023

**Study ID**: 16-1314


Study ID: 16-1314 Form Version Date: 6/29/2021

that contacting you is not practical, for example, because you have moved, your identifiable data and specimens may still be used. The Institutional Review Board (IRB) will be asked for permission to use the information and/or specimens linked to your identity. The IRB can give permission for researchers to use and share identifiable health information without contacting you, but only if it determines that sharing the information and/or specimens will not be more than a minimal risk to you or your privacy. The Institutional Review Board (IRB) is a committee of doctors and scientists and nonscientists, including people not associated with this hospital or medical school, whose job it is to protect people who participate in research.

| who participate | in research. |
|---|---|
| researchers, i | e permission to have portions of the specimens and/or information given <b>to other</b> ncluding those at Mount Sinai, other academic institutions and for profit companies, for a within the limits you have chosen above? Please initial your choice: |
| Yes | _ No |
| . , , . | e permission to have portions of the specimens and/or data <b>deposited in large public</b> (explained below) for use in research with the limits you may have chosen above? our choice: |
| Yes | _ No |
| numan sample<br>along with infor | werful research, it is helpful for researchers to share information they get from studying s. They do this by putting it into one or more scientific databases, where it is stored rmation from other studies. Researchers can then study the combined information to be about health and disease. If you agree to take part in this study, some of your |

To do more powerful research, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. Researchers can then study the combined information to learn even more about health and disease. If you agree to take part in this study, some of your genetic and health information might be placed into one or more scientific databases. There are many different kinds of scientific databases; some are maintained by Icahn School of Medicine at Mount Sinai or another institution, some are maintained by the federal government, and some are maintained by private companies. For example, the National Institutes of Health (an agency of the federal government) maintains a database called "dbGaP." A researcher who wants to study the information must apply for permission to use the database. Different databases may have different ways of reviewing such requests. Researchers with an approved study may be able to see and use your information, along with that from many other people. Researchers will always have a duty to protect your privacy and to keep your information confidential, but there are risks associated with data collection and sharing. They are described in more detail in the risks section.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study you will be responsible for the following things:

You would agree to undergo study procedures including follow-up visits, imaging, radical prostatectomy with permanent CivaSheet® implant and external beam radiation therapy.



#### ****

Study ID: 16-1314 Form Version Date: 6/29/2021

You would agree to fill out questionnaires before surgery and at each follow up visit after surgery requiring these questionnaires to be filled out.

You would agree to share relevant follow up clinical information when asked via mail or telephone when in person visits are not feasible for duration of 5 years after enrollment in the study.

### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for participating in this research study. Being in this research study will not lead to extra costs to you. You will not be reimbursed for your travel or time that may be required for study visits. The costs required for part of your standard of care will be your insurance's responsibility. The costs for the CivaSheet® will be covered by the study.

#### **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. While we hope that CivaSheet® with Radical Prostatectomy and Adjuvant External Beam Radiation Therapy will result in a reduced risk of cancer spread, a reduced risk of cancer recurrence and a reduced risk of death from prostate cancer, there is no evidence that this will occur. While we also hope that this combination treatment will reduce the unfavorable genitourinary and gastrointestinal effects of radiation to the bladder and rectum, there is no evidence that this will occur. Results from this trial may result in benefits to others. Determining the best dose of the CivaSheet® and whether this combination treatment is safe in this trial will allow us to safely treat future patients with the best dose of the CivaSheet® combined with radical prostatectomy and external beam radiation therapy to potentially reduce the risk of cancer spread, recurrence, death and complications related to radiation in other patients.

### REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:

The following information describes risks and side effects related to the procedures we are studying.

• This research involves two computed tomography scans. A computed tomography scan is a procedure relying on X-rays to obtain detailed intra-body images. A computed tomography scan often relies on a dye called contrast which may cause an allergic reaction (3%) such as nausea, vomiting, itching, sneezing hives or anaphylaxis (a life threatening allergic reaction) requiring intravenous medicines, intubation to allow breathing, or hospitalization which is rare. Other rare complications (0.04%) include loss of consciousness, cardiac arrest, difficult breathing (dyspnea) and low blood pressure (hypotension). Dye from computed tomography scans mwas say also damage your kidneys' function. A computed tomography scan will expose you to radiation which may increase your long term risk of developing cancer.



#### 


- This research involves blood tests to assess prostate specific antigen (PSA) levels and testosterone levels are part of follow-up visits. The risks of a blood draw include pain, bruising, and the slight possibility of infection at the place where the needle goes in. Some people feel dizzy or may faint during or after a blood draw.
- This research involves answering questionnaires at a pre-operative visit and at follow-up visits.
   Questionnaires are completed in the office and you may experience some psychological
   discomfort due to the personal nature of the questionnaires. Most patients do not feel bothered
   by such questions but there is always a potential risk for such an occurrence. You do not have
   to answer any questions you choose not to.
- This research involves radical prostatectomy (removal of the prostate and surrounding tissue). The rate of complications associated with robotic radical prostatectomy is 9% with only 2.42% major complications. Side effects related to radical prostatectomy will be monitored including but not limited to fever, chills, nausea, vomiting, abdominal pain, constipation, inability to urinate, blood in urine, blood in the stool, urine infection, sexual dysfunction (decreased erectile function), urine leak, lymphocele (a collection of lymph fluid needing to be drained), and death. Therefore, it is important to notify the research team of any symptoms or illness during the study period.
- This research involves external beam radiation therapy (delivery of high-energy x-rays to cancerous areas surrounding the prostate) following radical prostatectomy. Side effects related to external beam radiation therapy will also be monitored including but not limited to frequent urination, difficult or painful urination, blood in urine, urine leak, abdominal cramping, diarrhea, painful bowel movements, rectal bleeding, fatigue, sexual dysfunction including decreased erectile function and semen volume, skin reactions, secondary cancer resulting from radiation, urethral strictures, urinary incontinence, hematuria and lymphedema (fluid collection/swelling/pain in legs or genital region due to damage to lymph nodes around the prostate)
- In patients undergoing radical prostatectomy combined with external beam radiation therapy, common complications include urinary frequency (65.9%), diarrhea (61.3%), painful or difficult urination (49.2%), nausea or vomiting (4.4%), skin complications (38.3%), adverse bladder and rectal effects (21.9%), urethral stricture (17.8%), total urinary incontinence (6.5%), hematuria (4.6%) and rectal complications (rectal bleeding and inflammation) (3.3%).
- This research involves the permanent placement of Civasheet® in areas surrounding the prostate where cancer is known to have spread or is likely to have spread. CivaSheet® has not been used in any clinical trials to ascertain its risks or benefits. However, CivaSheet® is a low dose radiation sheet with palladium capsules on one side of the sheet and ¹o³palladium used in is often used for brachytherapy seed implantation which is known to result in the following complications: frequent urination which will affect 33% of men long term, urinary incontinence, urethral strictures, sexual dysfunction (decreased erectile function), rectal complications such as bleeding, pain, burning and diarrhea with serious long term complications occurring in less than 5% of patients. In patients with prostate cancer treated with 103 palladium brachytherapy




with or without external beam radiation therapy, common complications include acute urinary obstruction requiring a catheter (10-21%), rectal bleeding (5.6%) and impotency (39%). There may also be a risk of radiation to other areas due to movement of the Civasheet®. The Civasheet® will be sutured in place to minimize this risk. No studies have been conducted assessing the use of Civasheet® combined with radical prostatectomy and adjuvant external beam radiation therapy. We will therefore monitor side effects (e.g., fever, chills, infection, abscess, scarring, focal effects due to pressure like fistula, erosion into surrounding organs like perforation of viscera including bowel, bladder, bone, muscle, nerves and blood vessels) related to immune responses to immunologically foreign substances being placed in the body. The Civasheet® will be permanently implanted in you and emit internal radiation until the radiation is gone and the Civasheet® is no longer active. There may be a psychological risk in having the Civasheet® permanently inside your body. While this study is the first to assess the effectiveness and safety of Civasheet®, permanent placement of brachytherapy seeds consisting of 103 palladium (the same radiation source of the Civasheet®) are commonly used in the treatment of prostate, head/neck, cervical and breast cancer.

- Civasheet is a permanent brachytherapy device containing radiation. After 2 months, the radiation in the Civasheet will no longer be active. Since the radiation in the Civasheet will be active for 2 months, pregnant women and small children must not sit on your lap for 2 months.
  - There may also be side effects, other than listed above that we cannot predict. Most side effects go away shortly after the intervention is stopped.
  - Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

Combination therapy with radical prostatectomy, external beam radiation therapy and Civasheet® implant has never been assessed in the treatment of prostate cancer. Civasheet® has never been used in the treatment of prostate cancer. Therefore in addition to the stated risks above, this research may hurt you in ways that are not known. The unknown risks might be minor or might be major (death).

### OTHER POSSIBLE OPTIONS TO CONSIDER:

You may decide not to take part in this research study without any penalty. The choice is totally up to you.

Instead of being in this research study, your choices may include:

- Radical Prostatectomy with External Beam Radiation Therapy without the Civasheet.
- Radical Prostatectomy (Surgery to remove the prostate) alone.
- External Beam Radiation Therapy (delivery of high-energy x-rays to a patient's tumor or cancerous area) alone.



#### 


- Brachytherapy (a radioactive source such as palladium or iridium placed inside the tumor to destroy cancerous tissue) alone.
- Brachytherapy (a radioactive source such as palladium or iridium placed inside the tumor to destroy cancerous tissue) with external beam radiation therapy.
- Radical Prostatectomy with Hormonal Therapy.
- External Beam Radiation Therapy with Hormonal Therapy.

The important risks and possible benefits of these alternatives are listed below:

- Radical Prostatectomy with External Beam Radiation Therapy without the Civasheet.
  - Common complications for radical prostatectomy with external beam radiation therapy include urinary frequency (65.9%), diarrhea (61.3%), painful or difficult urination (49.2%), nausea or vomiting (4.4%), skin complications (38.3%), adverse bladder and rectal effects (21.9%), urethral stricture (17.8%), total urinary incontinence (6.5%), hematuria (4.6%) and rectal complications (rectal bleeding and inflammation) (3.3%).
  - Probability of death from any cause: 7-10%
- Radical Prostatectomy (Surgery to remove the prostate) alone.
  - The rate of complications associated with robotic radical prostatectomy is 9% with only 2.42% major complications. Side effects related to radical prostatectomy will be monitored including but not limited to fever, chills, nausea, vomiting, abdominal pain, constipation, inability to urinate, blood in urine, blood in the stool, urine infection, sexual dysfunction (decreased erectile function), urine leak, lymphocele (a collection of lymph fluid needing to be drained), and death. Therefore, it is important to notify the research team of any symptoms or illness during the study period.
  - Probability of death from any cause at 5 years: 8-12%
- External Beam Radiation Therapy (delivery of high-energy x-rays to a patient's tumor or cancerous area) alone.
  - Side effects related to external beam radiation therapy will also be monitored including but not limited to frequent urination, difficult or painful urination, blood in urine, urine leak, abdominal cramping, diarrhea, painful bowel movements, rectal bleeding, fatigue, sexual dysfunction including decreased erectile function and semen volume, skin reactions, secondary cancer resulting from radiation, urethral strictures, urinary incontinence, hematuria and lymphedema (fluid collection/swelling/pain in legs or genital region due to damage to lymph nodes around the prostate).
  - Probability of death from any cause at 5 years: 12.7%-15%
- External Beam Radiation Therapy with Hormonal Therapy
  - Side Effects within 3 months: Grade 1 gastrointestinal toxicity (51.67%) including anorexia with less than or equal to 5%, nausea, abdominal pain not requiring medication,




increased or changed bowel movements, and rectal discomfort. Grade 1 genitourinary toxicity (46.67%) including frequency of urination or nocturia two times per night, dysuria, and urinary urgency. Grade 2 gastrointestinal toxicity (44%) including anorexia with more than or equal to 15 % weight loss, nausea, rectal, abdominal pain and diarrhea requiring medication, mucous discharge not requiring sanitary pads. Grade 2 genitourinary toxicity (33.33%) including frequency or nocturia less frequent than every hour, dysuria, urgency and bladder spasms requiring local anesthesia. Grade 3 gastrointestinal toxicity (2.6%) including nausea, diarrhea or anorexia with > 15% weigh lost requiring nasogastric tube or parenteral support, severe abdominal pain even with medication, severe abdominal distension, severe mucous or blood discharge requiring sanitary pads, pneumonitis requiring intermittent oxygen or steroids. Grade 3 genitourinary toxicity (6.67%) including hourly or more frequent urination and nocturia, dysuria, pelvic pain, gross hematuria with or without clot passage and bladder spams requiring regular, frequent narcotics.

- Probability of death from any cause at 5 years: 7.7%-15%.
- Radical Prostatectomy with Hormonal Therapy
  - Side Effects: Miocardial infarction (2.2%), mild to moderate hematologic effects (15.2%), mild to moderate gastrointestinal effects (26.1%), mild to moderate incontinence (41.2%), urinary frequency (13%), nocturia (13%), hot flashes (50%), weight gain 17.4%), fatigue (4.3%), gynecomastia (21.7%) and severe hot flashes (8.7%). Severe abdominal pain, anxiety, cardiovascular events, rash, memory loss, hypertension and urinary changes may also occur (<3%),
  - Probability of death from any cause at 5 years: 4%-17.1%

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you are injured or made sick from taking part in this research study, medical care will be provided. Generally, this care will be billed to you or your insurance in the ordinary manner and you will be responsible for all treatment costs not covered by your insurance, including deductibles, co-payments and coinsurance. This does not prevent you from seeking payment for injury related to malpractice or negligence. Contact the investigator for more information

#### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

If you decide to stop being in the research study, please contact the Principal Investigator or the research staff.

If you decide to stop being in the research study, the following may occur you will continue to receive the standard of care which is radical prostatectomy with external beam radiation therapy.




If you stop being in the research study, already collected information may not be removed from the research study database and will continue to be used to complete the research analysis. You may be asked whether the investigator can collect information from your routine medical care. If you agree, this data will be handled the same as research data If you stop being in the study, no additional information will be collected.

You may also withdraw your permission for the use and disclosure of any of your protected information for research, but <u>you must do so in writing</u> to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from participating in the research study.

<u>Withdrawal without your consent</u>: The study doctor, the sponsor or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If data have been stored as part of the research study, they too can be destroyed without your consent. More possible reasons for removal from the study include spread of cancer to distant organs. If your cancer progresses and spreads to distant organs, you will be removed from the research and additional treatment options will be discussed such as hormone therapy, etc.

#### **CONTACT INFORMATION:**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Principal Investigator at 212-241-3919.

If you experience an emergency during your participation in this research, contact the Principal Investigator (Ketan Badani, MD) at phone number 212-241-3919, call 911, or go to the emergency room.

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.




| <b>Study ID</b> : 16-1314 | Form Version Date: 6/29/2021 |
|---------------------------|------------------------------|

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

The company (Civatech Oncology®) sponsoring this research study manufactures the drug/device being tested (Civasheet®) and so has a financial interest that could be affected by the outcome of this research study.

### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As you take part in this research project it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

What protected health information is collected and used in this study, and might also be disclosed (shared) with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, address, telephone/fax numbers, dates directly related to the individual (birth, admission, discharge, date of death, etc.), social security number, medical records number, health plan numbers, medical/surgical history, medications, laboratory/blood work results, procedural data, imaging data, data from questionnaires during office visits.

The researchers will also get information from your medical record from the Mount Sinai Hospital, Mount Sinai Hospital West and Mount Sinai St. Luke's Hospital.

During the study the researchers will gather information by:

- Taking a medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate and temperature
- Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.
- Reviewing HIV-related information, which includes any information indicating that you have had an HIV related test, or have HIV infection, HIV related illness or AIDS, or any information which could indicate that you have been potentially exposed to HIV




Why is your protected health information being used?

Your personal contact information is important to be able to contact you during the study. Your health information and the results of any tests and procedures being collected as part of this research study will be used for the purpose of this study as explained earlier in this consent form. The results of this study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The Principal Investigator may also use and share the results of these tests and procedures to treat you in collaboration with others in the Mount Sinai Health System.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

### Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator.)

- A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.
- The United States Department of Health and Human Services and the Office of Human Research Protection.
- Civatech Oncology, Inc.
- The United States Food and Drug Administration

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, the



### 


Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information?

Your authorization for use of your protected health information for this specific study does not expire.

Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The investigator is not required to release to you research information that is not part of your medical record.

Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

### Can you change your mind?

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your protected health information.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

• Your family members will not be contacted for clinical, research or other purposes without your consent.




If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is the case, the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may be ignored.

### Notice Concerning HIV-Related Information

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

IRB Approved


**Study ID**: 16-1314 Form Version Date: 6/29/2021 ADULT PARTICIPANT: Your signature below documents your permission to take part in this research and to the use and disclosure of your protected health information. A signed and dated copy will be given to you. Signature of subject Printed Name of Subject Date Time PERSON EXPLAINING STUDY AND OBTAINING CONSENT: Signature of consent delegate Printed Name of consent delegate Date Time WITNESS SECTION: When a witness is required to observe the consent process, it should be documented below (for example, when subject is illiterate, visually impaired, or this document accompanies a short form consent). My signature below documents that the information in the consent document and any other written information was accurately explained to, and apparently understood by, the subject, and that consent was freely given by the subject. Signature of Witness Printed Name of Witness Date Time

